CLINICAL TRIAL: NCT03332992
Title: Comparative Tests of Flu Vaccination Phone Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Emmi Solutions (Unknown); University of Iowa (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Brian Zikmund-Fisher, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00135995
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Health Insurance Portability and Accountability Act

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Viral changes + General intentions (Experimental): Script language discusses a) that previous years' shots do not protect against current year influenza (viral changes) and b) poses a general question asking whether the respondent intends to get a flu shot (general intentions).
  Interventions: Behavioral: Viral changes; Behavioral: General intentions
- Viral changes + Behavioral intentions (Experimental): Script language discusses a) that previous years' shots do not protect against current year influenza (viral changes) and b) poses a question asking when / where the respondent will get a flu shot (behavioral intention).
  Interventions: Behavioral: Viral changes; Behavioral: Behavioral intentions
- Viral changes + Accountability (Experimental): Script language discusses a) that previous years' shots do not protect against current year influenza (viral changes) and b) poses a question that implies the patient's care team will be notified of intent to vaccinate (accountability to providers).
  Interventions: Behavioral: Viral changes; Behavioral: Accountability
- Protect others + General intentions (Experimental): Script language discusses a) that getting the flu shot protects others who can get particularly sick (protect others) and b) poses a general question asking whether the respondent intends to get a flu shot (general intentions).
  Interventions: Behavioral: Protect others; Behavioral: General intentions
- Protect others + Behavioral intentions (Experimental): Script language discusses a) that getting the flu shot protects others who can get particularly sick (protect others) and b) poses a question asking when / where the respondent will get a flu shot (behavioral intention).
  Interventions: Behavioral: Protect others; Behavioral: Behavioral intentions
- Protect others + Accountability (Experimental): Script language discusses a) that getting the flu shot protects others who can get particularly sick (protect others) and b) poses a question that implies the patient's care team will be notified of intent to vaccinate (accountability to providers).
  Interventions: Behavioral: Protect others; Behavioral: Accountability

INTERVENTIONS:
Behavioral: Viral changes — Telephone script language provided pre-questions regarding the fact that influenza viruses change each year
  Arms: Viral changes + Accountability; Viral changes + Behavioral intentions; Viral changes + General intentions
Behavioral: Protect others — Telephone script language provided pre-questions emphasizing the need to protect vulnerable others
  Arms: Protect others + Accountability; Protect others + Behavioral intentions; Protect others + General intentions
Behavioral: General intentions — Question language asking about general interest in getting influenza vaccination
  Arms: Protect others + General intentions; Viral changes + General intentions
Behavioral: Behavioral intentions — Question language asking individual to make specific plans to be vaccinated
  Arms: Protect others + Behavioral intentions; Viral changes + Behavioral intentions
Behavioral: Accountability — Question language asking individual whether their care team can learn about their vaccination intentions
  Arms: Protect others + Accountability; Viral changes + Accountability

SUMMARY:
This project is a partnership between Emmi Solutions, a private company that delivers health promotion messages to employees of client organizations, and the University of Michigan and affiliated academic investigators. In particular, Emmi sends out pre-recorded and interactive telephone calls on behalf of their healthcare clients to promote influenza vaccination each Fall. The collaboration will design various scripts (based on established risk communication, behavior change, and behavioral economic principles) to be pre-recorded and sent out on these calls on a randomized basis (with approval by client organizations), with the number of arms to vary based on the size of each client's participant list (to ensure sufficient statistical power within each client's sample). Emmi will deliver the calls and track individual responses to questions posed during the call. Emmi will then provide a de-identified dataset to the academic research team for analysis to determine whether any scripts provided greater or lesser effects to people's their motivations to get a flu vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patient of client organizations of Emmi Solutions
* Provided a phone number to their care team

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7206 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Vaccination intentions (Time 1) | Day 1 (Assessed during the intervention telephone call)
  Question (language being manipulated) asking whether respondent intends to vaccinate

SECONDARY OUTCOMES:
Documented influenza vaccination | Within 6 months / during 2017-2018 influenza season
  Documentation (when available from Emmi Solutions' clients) via clients' employee records that influenza vaccination occurred

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Zikmund-Fisher, PhD, Principal Investigator — University of Michigan
Locations (1):
- Emmi Solutions, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03332992/Prot_SAP_000.pdf